CLINICAL TRIAL: NCT03626012
Title: A Phase 1 Multiple-Ascending-Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB078 Administered Intrathecally to Adults With C9ORF72-Associated Amyotrophic Lateral Sclerosis
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB078 in Adults With C9ORF72-Associated Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 245AS101; 2017-000294-36 (EudraCT Number)
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1: BIIB078 First Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB078
- Cohort 2: BIIB078 Second Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB078
- Cohort 3: BIIB078 Third Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by two maintenance doses on two later days.
  Interventions: Drug: BIIB078
- Cohort 4: BIIB078 Fourth Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: BIIB078
- Cohort 5: BIIB078 Fifth Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: BIIB078
- Cohort 6: BIIB078 Sixth Dosage (Experimental): BIIB078 will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by five maintenance doses on five later days.
  Interventions: Drug: BIIB078
- Cohorts 1-6: Placebo (Placebo Comparator): Matching placebo will be administered as a loading regimen of 3 doses, on Day 1 and two later days, followed by two maintenance doses on two later days (Cohorts 1 through 3) and five maintenance doses on five later days (Cohorts 4 through 6).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB078 — Administered as specified in the treatment arm.
  Arms: Cohort 1: BIIB078 First Dosage; Cohort 2: BIIB078 Second Dosage; Cohort 3: BIIB078 Third Dosage; Cohort 4: BIIB078 Fourth Dosage; Cohort 5: BIIB078 Fifth Dosage; Cohort 6: BIIB078 Sixth Dosage
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Cohorts 1-6: Placebo

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of BIIB078 in adults with C9ORF72-Amyotrophic Lateral Sclerosis (ALS). The secondary objectives of this study are to evaluate the pharmacokinetic profile of BIIB078 and to evaluate the effects of BIIB078 on clinical function. As the first-in-human study, the study enrolls a small number of participants in each cohort. Every participant in a cohort is treated with the same dose or placebo. The study is designed to evaluate and confirm the safety of each dose before enrolling and exposing new participants to a higher dose in the next cohort.

ELIGIBILITY:
Key Inclusion Criteria:

* Ability of the participant to understand the purpose and risks of the study, to provide signed and dated informed consent, and to authorize the use of confidential health information in accordance with national and local participant privacy regulations; or, in the event of the participant's physical incapacity to sign, to confirm that understanding and consent orally to a legally authorized representative (LAR) for the express purpose of having said informed consent and authorization signed on his/her behalf.
* All participants of childbearing potential must agree to practice highly effective contraception during the study and be willing and able to continue contraception for 5 months after their last dose of study treatment.
* Must meet the possible, laboratory-supported probable, probable, or definite criteria for diagnosing ALS according to the World Federation of Neurology El Escorial criteria and have documentation of a clinical genetic test demonstrating the presence of a pathogenic mutation in C9ORF72.
* Slow vital capacity (SVC) ≥ 50% of predicted value as adjusted for sex, age, and height (from the sitting position).
* Participants taking concomitant riluzole at study entry must be on a stable dose for ≥ 30 days prior to the first dose of study treatment (Day 1).
* Participants taking concomitant edaravone at study entry must be on a stable dose for ≥ 60 days prior to the first dose of study treatment (Day 1).
* ALS Cognitive Behavioral Screen (ALS-CBS) score ≥ 11 for the cognitive portion; ≥ 33 for the behavioral portion.
* Medically able to undergo the study procedures, and to adhere to the visit schedule at the time of study entry, as determined by the Investigator.
* Screening values of coagulation parameters including platelet count, international normalized ratio (INR), prothrombin time (PT), and activated partial thromboplastin time (APTT) should be within normal ranges.
* Has an informant/caregiver who, in the Investigator's judgment, has frequent and sufficient contact with the participant as to be able to provide accurate information about the participant's cognitive and functional abilities at Screening.

Key Exclusion Criteria:

* History of drug abuse or alcoholism ≤ 6 months of Screening that would limit participation in the study, as determined by the Investigator.
* Tracheostomy.
* Prescreening ALSFRS-R slope less than 0.4 points/month, where prescreening ALSFRS-R slope is defined as follows: (48 - ALSFRS-R score at Screening) / (months from date of symptom onset to date of Screening).
* History of or positive test result at Screening for human immunodeficiency virus. .
* History of, or positive test result at Screening for, hepatitis C virus antibody.
* Treatment with another investigational drug or biological agent within 1 month of Screening or 5 half-lives of study agent, whichever is longer.
* Treatment with an antiplatelet or anticoagulant therapy that cannot safely be interrupted for lumbar puncture (LP) according to local standard of care and/or institutional guidelines, in the opinion of the Investigator or Prescriber.
* Current or anticipated need, in the opinion of the Investigator, of a diaphragm pacing system during the study period.
* Female participants who are pregnant or currently breastfeeding.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline through End of Study (Approximately Day 323)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death, places participant at immediate risk of death, requires initial or prolonged inpatient hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly, is a medically important event.

SECONDARY OUTCOMES:
Serum BIIB078 Concentration | Baseline and at multiple time points up to Day 260
Area Under the Concentration-Time Curve (AUC) from Time 0 to Infinity (AUCinf) | Baseline and at multiple time points up to Day 260
AUC from Time 0 to Time of the Last Measurable Concentration (AUClast) | Baseline and at multiple time points up to Day 260
Maximum Observed Concentration (Cmax) | Baseline and at multiple time points up to Day 260
Time to Reach Cmax (Tmax) | Baseline and at multiple time points up to Day 260
Terminal Elimination Half-Life (t 1/2) | Baseline and at multiple time points up to Day 260
Change from Baseline in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) Scores | Baseline up to Day 323
  The ALSFRS-R has been demonstrated to predict survival. The ALSFRS-R measures 4 functional domains, including respiratory, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score of 48 [Cedarbaum 1999], with higher scores representing better function.
Change from Baseline in Percent of Predicted Slow Vital Capacity (SVC) | Baseline up to Day 260
Change from Baseline in Muscle Strength | Baseline up to Day 260
  Quantitative muscle strength will be evaluated using hand-held dynamometry (HHD), which tests isometric strength of multiple muscles using standard participant positioning. Approximately 8 muscle groups will be examined (per each side) in both upper and lower extremities.
Change from Baseline in Bulbar Strength | Baseline up to Day 260
  Bulbar strength will be measured by the Iowa Oral Pressure Instrument (IOPI). The IOPI is a commercially available tongue pressure measurement system composed of an air-filled bulb connected to a pressure transducer. The bulb can be placed in different positions in the mouth in order to assess different aspects of tongue weakness.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (21):
- United States (12):
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Palo Alto, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, New York, New York
  - Research Site, Knoxville, Tennessee
- Canada (3):
  - Research Site, Calgary, Alberta
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Research Site, Dublin, Ireland
- Research Site, Utrecht, Netherlands
- Research Site, Sankt Gallen, Switzerland
- United Kingdom (3):
  - Research Site, London, Greater London
  - Research Site, Sheffield, South Yorkshire
  - Research Site, London

REFERENCES:
- [Derived] van den Berg LH, Rothstein JD, Shaw PJ, Babu S, Benatar M, Bucelli RC, Genge A, Glass JD, Hardiman O, Libri V, Mobach T, Oskarsson B, Pattee GL, Ravits J, Shaw CE, Weber M, Zinman L, Jafar-Nejad P, Rigo F, Lin L, Ferguson TA, Gotter AL, Graham D, Monine M, Inra J, Sinks S, Eraly S, Garafalo S, Fradette S. Safety, tolerability, and pharmacokinetics of antisense oligonucleotide BIIB078 in adults with C9orf72-associated amyotrophic lateral sclerosis: a phase 1, randomised, double blinded, placebo-controlled, multiple ascending dose study. Lancet Neurol. 2024 Sep;23(9):901-912. doi: 10.1016/S1474-4422(24)00216-3. Epub 2024 Jul 23. PMID 39059407